CLINICAL TRIAL: NCT03085810
Title: An Open-Label, Single-Arm Study to Evaluate the Effectiveness and Safety of Ocrelizumab in Patients With Early Stage Relapsing Remitting Multiple Sclerosis
Brief Title: Study to Evaluate the Effectiveness and Safety of Ocrelizumab in Participants With Early Stage Relapsing Remitting Multiple Sclerosis (RRMS)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated earlier as the study sponsor collected sufficient data to perform all analyses as per pre-specified endpoints in the study protocol.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA30143; 2016-002937-31 (EudraCT Number)
Record Dates: First submitted 2017-03-16; First posted 2017-03-21 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ocrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ocrelizumab (Experimental): Ocrelizumab will be administered intravenously (IV) as two 300-milligram (mg) infusions (infusion length=2.5 hours) on Days 1 and 15, followed by one 600-mg infusion dose every 24 weeks (+/- 14 days) for a maximum of 8 doses throughout the 192 weeks treatment period.
  Interventions: Drug: Ocrelizumab
- Substudy Group 1 (Active Comparator): At week 24 of the main study, eligible participants will be randomized to receive 600 mg ocrelizumab infused over approximately 3.5 hours every 24 weeks for the remainder of the study duration
  Interventions: Drug: Ocrelizumab
- Substudy Group 2 (Experimental): At week 24 of the main study, eligible participants will be randomized to receive 600 mg ocrelizumab infused over approximately 2 hours followed by sodium chloride given as a slow infusion over the remaining 1.5 hours to mimic the standard-length infusion (3.5 hour) every 24 weeks for the remainder of the study duration
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab will be administered via IV infusion as specified throughout the treatment period.

SUMMARY:
This is a prospective, multicenter, open-label, single-arm, phase 3b study which evaluates effectiveness and safety of ocrelizumab in participants with early stage RRMS. The study will consist of an open-label treatment period of 192 weeks and follow-up period of at least 48 weeks.

The optional shorter infusion substudy will evaluate the safety of a shorter infusion of ocrelizumab in a subgroup of participants with early stage RRMS enrolled in the main MA30143 study. Approximately 700 patients will be enrolled in the substudy, and will receive additional 600 mg ocrelizumab administered in a shorter time frame.

ELIGIBILITY:
Inclusion Criteria:

* Have a definite diagnosis of RRMS, as per the revised McDonald 2010 criteria
* Have a length of disease duration, from first documented clinical attack consistent with MS disease of less than or equal to (</=) 3 years
* Within the last 12 months one or more clinically reported relapse(s) or one or more signs of MRI activity
* EDSS of 0.0 to 3.5 inclusive, at screening
* An agreement to use an acceptable birth control method for women of childbearing potential, during the treatment period and for at least 6 months or longer after the last dose of study drug

Exclusion Criteria:

* Secondary progressive multiple sclerosis or history of primary progressive or progressive relapsing MS
* Inability to complete an MRI
* Known presence of other neurological disorders

Exclusions Related to General Health:

* Pregnancy or lactation
* Participants intending to become pregnant during the study or within 6 months after the last dose of the study drug
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* History or currently active primary or secondary immunodeficiency
* Lack of peripheral venous access
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Significant or uncontrolled somatic disease or any other significant disease that may preclude participant from participating in the study
* Congestive heart failure (New York Heart Association III or IV functional severity)
* Known active bacterial, viral, fungal, mycobacterial infection or other infection, (excluding fungal infection of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks prior to screening or oral antibiotics 2 weeks prior to screening
* History of malignancy, major opportunistic infections, alcohol or drug abuse, recurrent or chronic infection, and/or coagulation disorders

Exclusions Related to Medications:

* Received any prior approved disease modifying treatment (DMT) with a label for MS, for example, interferons, glatiramer acetate, natalizumab, alemtuzumab, daclizumab, fingolimod, teiflunomide and dimethylfumarate
* Receipt of a live vaccine or attenuated live vaccine within 6 weeks prior to the baseline visit
* Previous treatment with B-cell targeted therapies (i.e., rituximab, ocrelizumab, atacicept, belimumab, or ofatumumab)
* Any previous treatment with immunosuppressants/ immunomodulators/ antineoplastic therapies (cyclophosphamide, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, cladribine, mitoxantrone, laquinimod, total body irradiation, or bone marrow transplantation)
* Treatment with investigational DMT
* Treatment with fampridine/dalfamipridine unless on stable dose for >/=30 days prior to screening

Exclusion related to Shorter Infusion Substudy:

- Any previous serious IRRs experienced with ocrelizumab treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1225 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (193):
- United States (26):
  - University of California Irvine, Irvine, California
  - Palo Alto Medical Foundation Research Center, Sunnyvale, California
  - University of Colorado Denver, Aurora, Colorado
  - Advanced Neurology of Colorado, LLC, Fort Collins, Colorado
  - KI Health Partners, LLC; New England Institute for Clinical Research, Stamford, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of South Florida - Bradenton, Tampa, Florida
  - Shepherd Center Inc., Atlanta, Georgia
  - College Park Family Care Ctr, Overland Park, Kansas
  - The NeuroMedical Center, Baton Rouge, Louisiana
  - Maine Medical Center, Scarborough, Maine
  - University of Maryland Medical Center; Department of Neurology, Baltimore, Maryland
  - Neurology Center of New England, Foxborough, Massachusetts
  - Dragonfly Research, LLC, Wellesley, Massachusetts
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Cleveland Clinic Lou Ruvo; Center for Brain Research, Las Vegas, Nevada
  - Columbia University Medical Center, New York, New York
  - Island Neurological Associates, P.C., Plainview, New York
  - Neurology Associates PA, Hickory, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation; Cleveland Clinic Cancer Center/I40, Cleveland, Ohio
  - Neurology Specialists, Inc, Dayton, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Kane Hall Barry Neurology, Bedford, Texas
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
  - Wheaton Franciscan Healthcare - St. Francis Outpatient Center; Center for Neurological Disorders, Milwaukee, Wisconsin
- Argentina (3):
  - Centro de Especialidades Neurológicas y Rehabilitación - CENyR, Buenos Aires
  - Hospital Churruca Visca, Buenos Aires
  - Fundacion Rosarina de Neurorehabilitacion, Rosario
- Australia (9):
  - Brain and Mind Centre, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Royal North Shore Hospital; Department of Neurology, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Box Hill Hospital; Department of Neurology, Box Hill, Victoria
  - Austin Hospital; Department of Neurology, Heidelberg, Victoria
  - Royal Melbourne Hospital; Department of Neurology, Parkville, Victoria
  - Perron Institute for Neurological and Translational Science, Nedlands, Western Australia
- Austria (4):
  - Medizinische Universität Graz; Universitätsklinik für Neurologie, Graz
  - Uniklinik fuer Neurologie, Medizinische Universitaet Innsbruck; Department fuer Neurologie, Innsbruck
  - Christian-Doppler-Klinik - Universitätsklinikum; Universitätskliniik für Neurologie, Salzburg
  - Medizinische Universität Wien; Univ.Klinik fuer Neurologie, Vienna
- Belgium (7):
  - AZ Sint Jan, Bruges
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - CHU Tivoli, La Louvière
  - CHU Sart-Tilman, Liège
  - Revalidatie en MS Centrum, Overpelt
- Brazil (4):
  - Hospital das Clinicas - UFMG, Belo Horizonte, Minas Gerais
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - FMUSP, São Paulo, São Paulo
- Bulgaria (3):
  - Shat Np Sveti Naum; 3Rd Clinic of Neurology, Sofia
  - Multiprofile Hosp. for Active Treatment;National Cardiology Hosp., Sofia
  - UMHAT Alexandrovska, EAD; Neurology, Sofia
- Canada (7):
  - UBC Hospital; Div of Neurology, Dept of Medicine, Vancouver, British Columbia
  - London Health Sciences Centre Uni Campus, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Clinique NeuroOutaouais, Gatineau, Quebec
  - Recherche Sepmus Inc., Greenfield Park, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- Denmark (3):
  - Aalborg Universitetshospital; Neurologisk Afdeling og Neurofysiologisk Afdeling; Skleroseamb., Aalborg
  - Aarhus Universitetshospital; Neurologisk Afd. F, Skleroseklinikken, Aarhus N
  - Rigshospitalet; Neurologisk Klinik Glostrup, Glostrup Municipality
- France (20):
  - CHU de Besancon Hopital Jean Minjoz; Service de Neurologie, Besançon
  - Hopital Pellegrin-CHU de Bordeaux; Service de Neurologie, Bordeaux
  - Hopital Pierre Wertheimer; Neurologie D, Bron
  - CHU de Caen Hopital Cote de Nacre, Caen
  - CHU Hopital Gabriel Montpied; Service de Neurologie, Clermont-Ferrand
  - CH de Gonesse; Neurologie, Gonesse
  - CHU de Grenoble; Neurologie, La Tronche
  - Hopital Gui de Chauliac; Neurologie, Montpellier
  - Hopital Central - CHU de Nancy; Service de Neurologie, Nancy
  - Hôpital Guillaume et René Laënnec; Service Neurologie, Nantes
  - Hôpital Pasteur; Service de Neurologie, Nice
  - CHU de Nîmes Hopital Caremeau; Service de Neurologie, Nîmes
  - Hôpital de Poissy; Service neurologie, Poissy
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - CHU de Rouen Hopital; Service de Neurologie, Rouen
  - CHU de Strasbourg, Strasbourg
  - Hopital Foch; Neurologie, Suresnes
  - HIA de Toulon hôpital militaire; Neurologie, Toulon
  - CHU toulouse - Hôpital Purpan; Departement de Neurologie, Toulouse
  - CHRU - Hôpital Bretonneau; Neurologie, Tours
- Germany (18):
  - Praxis Dr.med. Sylvia Menck, Fachärztin für Neurologie und Psychiatrie, Barsinghausen
  - Jüdisches Krankenhaus Berlin; Abteilung fur Neurologie, Berlin
  - St. Josef-Hospital, Klinik für Neurologie, Bochum
  - Studienzentrum Dr. Bischof GmbH, Böblingen
  - Universitätsklinikum "Carl Gustav Carus", Zentrum für Klinische Neurowissenschaften, Dresden
  - Universitätsklinikum Düsseldorf; Klinik für Neurologie, Düsseldorf
  - NeuroCentrum Odenwald; Dres. Reifschneider, Unsorg, Ries, Schumann, Hoffmann, Knoblich, Erbach/Odenwald
  - Universitätsklinikum Essen (AöR); Klinik für Neurologie, Essen
  - MultipEL Studies - Institut für klinische Studien, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Neurologische Gemeinschaftspraxis Kassel und Vellmar, Ch. Lassek, Dres. Ammerbach, Fetzer, M. Fische, Kassel
  - Uniklinik Schleswig-Holstein; Neuroimmunologie, Institut für Klinische Chemie + Klinik f. Neurologie, Kiel
  - Universitaetsklinikum Marburg; Klinik fuer Neurologie, Marburg
  - Klinikum rechts der Isar der TU Muenchen; Neurologische Klinik und Poliklinik im Neuro-Kopf-Zentrum, München
  - Universitätsklinikum Münster; Klinik und Poliklinik für Neurologie, Münster
  - Praxis Dr. med. Bergmann, Neuburg am Inn
  - Asklepios Kliniken Schildautal Seesen; Klinik für Neurologie, Seesen
  - Universitätsklinikum Tübingen, Zentrum für Neurologie, Tübingen
- Hungary (5):
  - Semmelweis Egyetem AOK; Neurologiai Klinika, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
  - Jahn Ferenc Dél-Pesti Kórház, Budapest
  - VALEOMED Diagnosztikai Központ, Esztergom
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ; Neurológiai Klinika, Szeged
- Italy (16):
  - A.O.U. Mater Domin; U.O. NEUROLOGIA, Catanzaro, Calabria
  - A. O. U. Federico II; Dip Neuroscienze, Scienze Riproduttive ed Odontostomatologiche, Napoli, Campania
  - Università degli Studi della Campania Luigi Vanvitelli; Dip. Ass. Integrato Med Int-II Clinica Neur, Napoli, Campania
  - Ospedale Cattinara; Amb Studio Sclerosi Multipla, Clinica Neurlogica, Trieste, Friuli Venezia Giulia
  - Policlinico Tor Vergata Dip. Neuroscienze-Clinica Neurologica-UOSD Sclerosi Multipla, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea; UOC Neurologia, Rome, Lazio
  - Irccs A.O.U.San Martino Ist; Dinogmi, Genoa, Liguria
  - IRCCS Ospedale San Raffaele; Neurologia Neurofisiologia Neuroriabilitazione-Centro Sclerosi Multipla, Milan, Lombardy
  - Fond. Istituto Neurologico C.Besta; UO Neurologia IV - Neuroimmunologia Malattie Neuromuscolari, Milan, Lombardy
  - Ospedale Civile di Montichiari; Centro Sclerosi Multipla, Montichiari, Lombardy
  - IRCCS Istituto Neurologico Neuromed; Centro per lo Studio e la Cura della Sclerosi Multipla, Pozzilli, Molise
  - AOU Policlinico V. Emanuele - P.O G. Rodolico; Clinica Neurologica, Centro Sclerosi Multipla, Catania, Sicily
  - AO Ospedali Riuniti Villa Sofia-Cervello;PO Villa Sofia - UO Neurologia - U.O.S. Neuroimmunologia, Palermo, Sicily
  - AOU Careggi; Neurologia 1-Dip. Neuroscienze Psicologia Area Farmaco Salute del Bambino(NEUROFARBA), Florence, Tuscany
  - Ospedale Misericordia USL9 di Grosseto; U.O. Neurologia, Grosseto, Tuscany
  - Ospedale Le Scotte; Clinica Neurologica e Malattie Neurometaboliche, Siena, Tuscany
- Ibn Sina Hospital; Neurology Department, Kuwait City, Kuwait
- American University of Beirut - Medical Center, Beirut, Lebanon
- Mexico (3):
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
  - Hospital General de Mexico, Mexico, Tlaxcala
  - Unidad de investigacion en salud (UIS); Neurociencias, Mexico City
- Netherlands (4):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - VU Medisch Centrum; Afdeling Neurologie, Amsterdam
  - Groene Hart Ziekenhuis, Gouda
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
- Norway (2):
  - Akershus universitetssykehus HF; Nevroklinikken S203, Lørenskog
  - Stavanger Universitetssykehus, Helse Stavanger HF, Stavanger
- Poland (8):
  - Neurocentrum Bydgoszcz sp. z o.o, Bydgoszcz
  - COPERNICUS Podmiot Leczniczy Sp. z o. o. Szpital im. M. Kopernika; Oddzia? Neurologiczny, Gdansk
  - Care Clinic, Katowice
  - Malopolskie Centrum Diagnostyczne MEDICAL Sp. z o. o., Krakow
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Indywidualna Praktyka Lekarska Prof. Dr Hab. N. Med. Konrad Rejdak., Lublin
  - Klinika Neurologii I Wydzialu Lekarskiego WUM w Warszawie, Warsaw
  - Instytut Psychiatrii i Neurologii II Klinika Neurologiczna, Warsaw
- Portugal (5):
  - Hospital Garcia de Orta; Servico de Neurologia, Almada
  - Hospital de Braga; Servico de Neurologia, Braga
  - HUC; Servico de Neurologia, Coimbra
  - Hospital Beatriz Angelo; Servico de Neurologia, Loures
  - Hospital Geral de Santo Antonio; Servico de Neurologia, Porto
- Romania (3):
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Clinic Judetean Sibiu, Sibiu
  - Spitalul Clinic Judetean de Urgenta Mures, Târgu Mureş
- Slovakia (4):
  - Univerzitna nemocnica Bratislava, Nemocnica Staré Mesto; I. Neurologická klinika SZU a UNB, Bratislava
  - Univerzitna nemocnica Bratislava - Nemocnica Ruzinov; Neurologicka klinika SZU a UNB, Bratislava
  - GB NeuroPRAKTIK, s.r.o, Nitra
  - Fakultna nemocnica Trnava, Trnava
- Slovenia (2):
  - University Medical Centre; Neurology, Ljubljana
  - University Medical Centre Maribor, Maribor
- Spain (7):
  - Complejo Hospitalario Nuestra Señora de la Candelaria; Servicio de Neurologia, Santa Cruz de Tenerife, Tenerife
  - Hospital de Cruces; Servicio de Neurologia, Barakaldo, Vizcaya
  - Hospital General Universitario de Alicante; Servicio de Neurología, Alicante
  - Hospital del Mar; Servicio de Neurologia, Barcelona
  - Hospital Vall d'Hebron; Servicio de Neurología, Barcelona
  - Hospital Universitario Puerta De Hierro Majadahonda; Servicio de Neurología, Madrid
  - Hospital General Universitario Morales Meseguer; Servicio de Neurología, Murcia
- Sweden (3):
  - Sahlgrenska Sjukhuset; Neurology, Gothenburg
  - Centralsjukhuset; Neurologi och rehabiliteringskliniken, Karlstad
  - Centrum för Neurologi, Stockholm
- Switzerland (5):
  - Universitätsspital Basel; Neurologie, Basel
  - Inselspital Bern Medizin Neurologie; Neurologische Poliklinik, Bern
  - Luzerner Kantonsspital Luzern Medizin Neurologie, Lucerne
  - Ospedale Regionale di Lugano - Civico; Neurologia, Lugano
  - Kantonsspital; Neurologische Klinik, Sankt Gallen
- Turkey (Türkiye) (9):
  - Hacettepe University Medical Faculty; Neurology, Ankara
  - Gazi University Medical Faculty; Departmant of Norology, Ankara
  - Mustafa Kemal Ataturk UTF; Department of norology, Hatay
  - Istanbul University Istanbul Medical Faculty; Neurology, Istanbul
  - Istanbul Universitesi - Cerrahpasa Cerrahpasa Tip Fakultesi; Noroloji Anabilim Dali, Istanbul
  - Istanbul Bilim Universty Medical Fac., Istanbul
  - Selcuk University Medical Faculty; Norology department, Istanbul
  - Ondokuz Mayis Univ. Med. Fac.; Neurology, Samsun
  - Karadeniz Tecnical Uni. Med. Fac.; Neurology, Trabzon
- United Kingdom (10):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Queen Elizabeth University Hospital, Glasgow
  - Royal Free Hospital, London
  - King'S College Hospital, London
  - Charing Cross Hospital, London
  - National Hospital for Neurology and Neurosurgery,; MRC Centre for Neuromuscular Diseases, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Derriford Hospital, Plymouth
  - Salford Royal NHS Foundation Trust, Salford
  - Abertawe and Bro Morgannwg NHS Trust; Clinical Researdh Institute, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Kappos L, Yiu S, Reucassel J, Oh J, Granziera C, Killestein J, Bermel RA, Berge C, Kazlauskaite A, Schneble HM, Dahlke F, Cree BAC. Performance of Composite Endpoints Defining Progression Independent of Relapse Activity in Multiple Sclerosis. Ann Clin Transl Neurol. 2025 Sep;12(9):1805-1812. doi: 10.1002/acn3.70111. Epub 2025 Jul 8. PMID 40629721
- [Derived] Kappos L, Yiu S, Dahlke F, Coetzee T, Cutter GR, Yuen S, Bonati U, Lublin FD. Composite Confirmed Disability Worsening/Progression Is a Useful Clinical Endpoint for Multiple Sclerosis Clinical Trials. Neurology. 2025 May 27;104(10):e213558. doi: 10.1212/WNL.0000000000213558. Epub 2025 Apr 21. PMID 40258203
- [Derived] Hartung HP, Benedict RHB, Berger T, Bermel RA, Brochet B, Carroll WM, Freedman MS, Holmoy T, Karabudak R, Nos C, Patti F, Perrin Ross A, Vanopdenbosch L, Vollmer T, Wuerfel J, Clinch S, Kadner K, Kuenzel T, Kulyk I, Raposo C, Thanei GA, Killestein J. Ocrelizumab in Early-Stage Relapsing-Remitting Multiple Sclerosis: The Phase IIIb ENSEMBLE 4-Year, Single-Arm, Open-Label Trial. Neurology. 2024 Dec 24;103(12):e210049. doi: 10.1212/WNL.0000000000210049. Epub 2024 Dec 3. PMID 39626127
- [Derived] Hartung HP, Berger T, Bermel RA, Brochet B, Carroll WM, Holmoy T, Karabudak R, Killestein J, Nos C, Patti F, Perrin Ross A, Vanopdenbosch L, Vollmer T, Buffels R, Garas M, Kadner K, Manfrini M, Wang Q, Freedman MS. ENSEMBLE PLUS: final results of shorter ocrelizumab infusion from a randomized controlled trial. J Neurol. 2024 Jul;271(7):4348-4360. doi: 10.1007/s00415-024-12326-z. Epub 2024 Apr 22. PMID 38649522
- [Derived] Hartung HP; ENSEMBLE Steering Committee members and study investigators. Ocrelizumab shorter infusion: Primary results from the ENSEMBLE PLUS substudy in patients with MS. Neurol Neuroimmunol Neuroinflamm. 2020 Jun 4;7(5):e807. doi: 10.1212/NXI.0000000000000807. Print 2020 Sep. PMID 32503093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A prospective, multicenter, open-label, single-arm effectiveness and safety study enrolled 1225 eligible treatment-naive patients with early stage RMSR. The study consisted of screening period up 4 weeks and open-label treatment with ocrelizumab period up to 192 week.
Pre-assignment Details: The efficacy analyses were performed on the main study cohort enrolled as per original study protocol, and safety analyses on all enrolled participants.
Groups:
- Main Study - Ocrelizumab: Ocrelizumab was administered intravenously (IV) as two 300-milligram (mg) infusions on Days 1 and 15, followed by one 600-mg infusion dose every 24 weeks (+/- 14 days) for a maximum of 8 doses throughout the 192 weeks treatment period.
- Substudy - Conventional Infusion: Ocrelizumab was administered as 600 mg IV infused over approximately 3.5 hours every 24 weeks throughout the treatment period.
- Substudy - Shorter Infusion: Ocrelizumab was administered as 600 mg IV infused over approximately 2 hours and saline for remaining 1.5 hours, every 24 weeks throughout the treatment period.
Period: Main Study
Arm/Group | Main Study - Ocrelizumab | Substudy - Conventional Infusion | Substudy - Shorter Infusion
Started | 1225 | 0 | 0
Completed | 1010 | 0 | 0
Not Completed | 215 | 0 | 0
Not completed — Withdrawal by Subject | 77 | 0 | 0
Not completed — Terminated By Sponsor | 14 | 0 | 0
Not completed — Protocol Violation | 15 | 0 | 0
Not completed — Physician Decision | 13 | 0 | 0
Not completed — Lost to Follow-up | 17 | 0 | 0
Not completed — Adverse Event | 25 | 0 | 0
Not completed — Pregnancy | 7 | 0 | 0
Not completed — Changed to Commercial Ocrelizumab | 4 | 0 | 0
Not completed — Lack of Efficacy | 10 | 0 | 0
Not completed — Death | 12 | 0 | 0
Not completed — Disease progression | 1 | 0 | 0
Not completed — Site Closure | 3 | 0 | 0
Not completed — Planned pregnancy | 17 | 0 | 0
Period: Substudy (Week 24 to Week 144)
Arm/Group | Main Study - Ocrelizumab | Substudy - Conventional Infusion | Substudy - Shorter Infusion
Started | 0 | 373 | 372
Completed | 0 | 0 | 2
Not Completed | 0 | 373 | 370
Not completed — Withdrawal due to Infusion Related Reaction (IRR) | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 5 | 7
Not completed — Substudy Stopped by Sponsor | 0 | 355 | 352
Not completed — Reason Not Specified | 0 | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Ocrelizumab: Ocrelizumab was administered intravenously (IV) as two 300-milligram (mg) infusions on Days 1 and 15, followed by one 600-mg infusion dose every 24 weeks (+/- 14 days) for a maximum of 8 doses throughout the 192 weeks treatment period
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 1225
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 784
  Male | 441
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 145
  Not Hispanic or Latino | 960
  Unknown or Not Reported | 120
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 34
  White | 1007
  More than one race | 37
  Unknown or Not Reported | 115

OUTCOME MEASURES:

1. Primary Outcome: Time to Onset of Confirmed Disability Progression (CDP) Sustained for at Least 24 Weeks and 48 Weeks as Measured Using Expanded Disability Status Scale (EDSS)
Description: The EDSS-Expanded Disability Status Scale is a disability scale that ranges in 0.5-point steps from 0 (normal) to 10 (death). Disability progression as measured by EDSS is defined as ≥1 point increase in EDSS score from a baseline EDSS score of 1-5 inclusive, a 0.5-increase from a baseline EDSS score higher than 5 and a 1.5-increase from a baseline EDSS score from 0 to 1 exclusive. Disability progression was considered confirmed if a sustained change in EDSS for a minimum of 24 weeks (-2 weeks) from the initial progression event was seen i.e. the change in EDSS must have been sustained at all available visits for a minimum of 24 weeks/48 weeks.
Time Frame: Baseline up to 4 years
Population: Treatment efficacy was measured for this First Enrollment Cohort ITT population.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Ocrelizumab: First Enrollment Cohort. Ocrelizumab was administered intravenously (IV) as two 300-milligram (mg) infusions on Days 1 and 15, followed by one 600-mg infusion dose every 24 weeks (+/- 14 days) for a maximum of 8 doses throughout the 192 weeks treatment period
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
weeks
  CPD Sustained for at Least 24 weeks | NA [NA to NA] — Median (corresponds to a probability of 50%) and 95% CI was not reached due to low number of participants with the event at the end of the study.
  CDP Sustained for at Least 48 weeks | NA [NA to NA] — Median (corresponds to a probability of 50%) and 95% CI was not reached due to low number of participants with the event at the end of the study.

2. Primary Outcome: Percentage of Participants With 24-Week and 48-Week Confirmed Disability Improvement (CDI) During the Year 1 Treatment Period, as Measured Using EDSS
Description: CDI is defined as an improvement of ≥1 point on the EDSS score confirmed at a regular scheduled visit at least 24/48 weeks after the initial documentation of neurological worsening (measured only participants with a baseline EDSS of ≥2.0). EDSS is a disability scale that ranges in 0.5-point steps from 0 (normal) to 10 (death).
Time Frame: At Weeks 24 and 48 during Year 1
Population: Treatment efficacy was measured for this First Enrollment Cohort ITT population. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses at the specified timepoints.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 309
Percentage of Participants
  CDI Sustained for 24 weeks: At Week 24: number analyzed (Participants) | 293
  CDI Sustained for 24 weeks: At Week 24 | 95.11 [92.03 to 97.03]
  CDI Sustained for 24 weeks: At Week 48: number analyzed (Participants) | 205
  CDI Sustained for 24 weeks: At Week 48 | 83.50 [78.81 to 87.24]
  CDI Sustained for 48 weeks: At Week 48: number analyzed (Participants) | 213
  CDI Sustained for 48 weeks: At Week 48 | 87.54 [83.28 to 90.77]

3. Primary Outcome: Percentage of Participants Event-Free for CDP Sustained for at Least 24 and 48 Weeks at Year 1, as Measured Using EDSS
Description: The EDSS-Expanded Disability Status Scale is a disability scale that ranges in 0.5-point steps from 0 (normal) to 10 (death). Disability progression as measured by EDSS is defined as ≥1 point increase in EDSS score from a baseline EDSS score of 1-5 inclusive, a 0.5-increase from a baseline EDSS score higher than 5 and a 1.5-increase from a baseline EDSS score from 0 to 1 exclusive. Disability progression was considered confirmed if a sustained change in EDSS for a minimum of 24 weeks (-2 weeks) from the initial progression event was seen i.e. the change in EDSS must have been sustained at all available visits (during Year 1) for a minimum of 24 weeks/48 weeks. Percentage of participants who did not have CPD sustained for 24 and 48 weeks are reported here.
Time Frame: Year 1 (Weeks 24 and 48)
Population: Treatment efficacy was measured for this First Enrollment Cohort ITT population. Number analyzed per timepoint are unique number of participants out of all the participants who were assessed for CDP at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage of Participants
  CDP Sustained for 24 weeks: At Week 24: number analyzed (Participants) | 668
  CDP Sustained for 24 weeks: At Week 24 | 99.55 [98.62 to 99.86]
  CDP Sustained for 24 weeks: At Week 48: number analyzed (Participants) | 645
  CDP Sustained for 24 weeks: At Week 48 | 97.30 [95.75 to 98.29]
  CDP Sustained for 48 weeks: At Week 48: number analyzed (Participants) | 649
  CDP Sustained for 48 weeks: At Week 48 | 98.05 [96.67 to 98.87]

4. Primary Outcome: Percentage of Participants With 24-Week and 48-Week CDI During the Year 2 Treatment Period, as Measured Using EDSS
Description: CDI is defined as an improvement of 1 point on the EDSS score confirmed at a regular scheduled visit at least 24/48 weeks after the initial documentation of neurological worsening (measured only participants with a baseline EDSS of ≥2.0). EDSS is a disability scale that ranges in 0.5-point steps from 0 (normal) to 10 (death).
Time Frame: At Weeks 48, 72 and 96 during Year 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 252
Percentage of Participants
  CDI Sustained for 24 weeks: At Week 48 | 100.0 [100.00 to 100.00]
  CDI Sustained for 48 weeks: At Week 48 | 100.00 [100.00 to 100.00]
  CDI Sustained for 24 weeks: At Week 72:: number analyzed (Participants) | 243
  CDI Sustained for 24 weeks: At Week 72: | 97.20 [94.22 to 98.66]
  CDI Sustained for 48 weeks: At Week 72: number analyzed (Participants) | 244
  CDI Sustained for 48 weeks: At Week 72 | 97.60 [94.74 to 98.91]
  CDI Sustained for 24 weeks: At Week 96: number analyzed (Participants) | 166
  CDI Sustained for 24 weeks: At Week 96 | 90.29 [85.71 to 93.46]
  CDI Sustained for 48 weeks: At Week 96: number analyzed (Participants) | 169
  CDI Sustained for 48 weeks: At Week 96 | 92.55 [88.41 to 92.55]

5. Primary Outcome: Percentage of Participants Event-free for CDP Sustained for at Least 24 and 48 Weeks at Year 2, as Measured Using EDSS
Description: as for outcome 3
Time Frame: Year 2 (Weeks 72 and 96)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Particiopants
Groups:
- Ocrelizumab: Ocrelizumab was administered intravenously (IV) as two 300-milligram (mg) infusions (infusion length=2.5 hours) on Days 1 and 15, followed by one 600-mg infusion dose every 24 weeks (+/- 14 days) for a maximum of 8 doses throughout the 192 weeks treatment period
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage of Particiopants
  CDP Sustained for 24 weeks: At Week 72: number analyzed (Participants) | 615
  CDP Sustained for 24 weeks: At Week 72 | 93.97 [91.87 to 95.54]
  CDP Sustained for 48 weeks: At Week 72: number analyzed (Participants) | 622
  CDP Sustained for 48 weeks: At Week 72 | 95.18 [93.25 to 96.56]
  CDP Sustained for 24 weeks: Week 96: number analyzed (Participants) | 587
  CDP Sustained for 24 weeks: Week 96 | 91.65 [89.26 to 93.52]
  CDP Sustained for 48 weeks: Week 96: number analyzed (Participants) | 598
  CDP Sustained for 48 weeks: Week 96 | 93.47 [91.30 to 95.12]

6. Primary Outcome: Percentage of Participants With 24-Week and 48-Week CDI at Year 4, as Measured Using EDSS
Description: CDI is defined as an improvement of 1 point on the EDSS score confirmed at a regular scheduled visit at least 24 weeks after the initial documentation of neurological worsening (measured only participants with a baseline EDSS of ≥2.0). EDSS is a disability scale that ranges in 0.5-point steps from 0 (normal) to 10 (death).
Time Frame: At Weeks 144, 168 and 192 during Year 4
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage of Participants
  CDI Sustained for 24 weeks: At Week 144: number analyzed (Participants) | 218
  CDI Sustained for 24 weeks: At Week 144 | 100.00 [100.00 to 100.00]
  CDI Sustained for 48 weeks: At Week 144: number analyzed (Participants) | 218
  CDI Sustained for 48 weeks: At Week 144 | 100.00 [100.00 to 100.00]
  CDI Sustained for 24 weeks: At Week 168: number analyzed (Participants) | 215
  CDI Sustained for 24 weeks: At Week 168 | 99.54 [96.77 to 99.93]
  CDI Sustained for 48 weeks: At Week 168: number analyzed (Participants) | 216
  CDI Sustained for 48 weeks: At Week 168 | 100.00 [100.00 to 100.00]
  CDI Sustained for 24 weeks: At Week 192: number analyzed (Participants) | 163
  CDI Sustained for 24 weeks: At Week 192 | 93.77 [89.51 to 96.34]
  CDI Sustained for 48 weeks: At Week 192: number analyzed (Participants) | 172
  CDI Sustained for 48 weeks: At Week 192 | 98.01 [94.77 to 99.25]

7. Primary Outcome: Percentage of Participants Event-free for CDP Sustained for at Least 24 and 48 Weeks at Year 4, as Measured Using EDSS
Description: as for outcome 3
Time Frame: Year 4 (Weeks 168 and 192)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage of Participants
  CDP Sustained for 24 weeks: At Week 168: number analyzed (Participants) | 516
  CDP Sustained for 24 weeks: At Week 168 | 85.98 [83.04 to 88.44]
  CDP Sustained for 48 weeks: At Week 168: number analyzed (Participants) | 528
  CDP Sustained for 48 weeks: At Week 168 | 87.98 [85.20 to 90.27]
  CDP Sustained for 24 weeks: At Week 192: number analyzed (Participants) | 402
  CDP Sustained for 24 weeks: At Week 192 | 84.18 [81.08 to 86.81]
  CDP Sustained for 48 weeks: At Week 192: number analyzed (Participants) | 414
  CDP Sustained for 48 weeks: At Week 192 | 86.48 [83.54 to 88.93]

8. Primary Outcome: Percentage of Participants Who Have Improved, Stable, or Worsened Disability Compared to Baseline at Year 1, As Measured Using EDSS
Time Frame: Year 1 (Week 48)
Population: First Enrollment Cohort ITT population. Treatment efficacy was measured for this First Enrollment Cohort. Overall number analyzed is the number of participants with data available for analyses.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 659
Percentage of Participants
  Week 48 Worsened (>0.5) | 9.3
  Week 48 Stable (Change <= 0.5 and >= -0.5) | 73.3
  Week 48 Improved (<-0.5) | 17.5

9. Primary Outcome: Percentage of Participants Who Have Improved, Stable, or Worsened Disability Compared to Baseline at Year 2, As Measured Using EDSS
Time Frame: Year 2 (Week 96)
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 632
Percentage of Participants
  Week 96 Worsened (>0.5) | 11.9
  Week 96 Stable (Change <= 0.5 and >= -0.5) | 76.6
  Week 96 Improved (<-0.5) | 11.6

10. Primary Outcome: Percentage of Participants Who Have Improved, Stable, or Worsened Disability at Year 3, As Measured Using EDSS
Time Frame: Year 3
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 557
Percentage of Participants
  Worsened (>0.5) | 9.3
  Stable (Change <= 0.5 and >= -0.5) | 81.5
  Improved (<-0.5) | 9.2

11. Primary Outcome: Percentage of Participants Who Have Improved, Stable, or Worsened Disability at Year 4, As Measured Using EDSS
Time Frame: Year 4
Population: as for outcome 8
Measure: Number; unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 562
Percentage of Participants
  Worsened (>0.5) | 18.0
  Stable (Change <= 0.5 and >= -0.5) | 59.3
  Improved (<-0.5) | 22.8

12. Primary Outcome: Mean Change From Baseline in EDSS Score at Week 24
Time Frame: From Baseline to Week 24
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Change in Total EDSS Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 671
Change in Total EDSS Score | -0.14 (0.68)

13. Primary Outcome: Mean Change From Baseline in EDSS Score at Week 48
Time Frame: From Baseline to Week 48
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Change in Total EDSS Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 659
Change in Total EDSS Score | -0.14 (0.77)

14. Primary Outcome: Mean Change From Baseline in EDSS Score at Week 72
Time Frame: From Baseline to Week 72
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Change in Total EDSS Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 651
Change in Total EDSS Score | -0.09 (0.89)

15. Primary Outcome: Mean Change From Baseline in EDSS Score at Week 96
Time Frame: Baseline, Week 96
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Change in Total EDSS Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 637
Change in Total EDSS Score | -0.12 (0.95)

16. Primary Outcome: Mean Change From Baseline in EDSS Score at Week 120
Time Frame: Baseline, Week 120
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Change in Total EDSS Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 579
Change in Total EDSS Score | -0.10 (0.94)

17. Primary Outcome: Mean Change From Baseline in EDSS Score at Week 144
Time Frame: Baseline, Week 144
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Change in Total EDSS Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 561
Change in Total EDSS Score | -0.10 (1.00)

18. Primary Outcome: Mean Change From Baseline in EDSS Score at Week 168
Time Frame: Baseline, Week 168
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Change in Total EDSS Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 560
Change in Total EDSS Score | -0.05 (1.05)

19. Primary Outcome: Mean Change From Baseline in EDSS Score at Week 192
Time Frame: Baseline, Week 192
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Change in Total EDSS Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 562
Change in Total EDSS Score | -0.06 (1.06)

20. Primary Outcome: Percentage of Participants Without Protocol-Defined Event of Disease Activity
Description: Protocol-defined event of disease activity is defined as having at least one of the following: (1). protocol defined relapse (occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis [MS], as determined using EDSS/Functional Systems Score [FSS] assessment). (2). CDP, as determined using EDSS. (3). a T1 Gd-enhanced lesion after Week 8 (4). a new and/or enlarging T2 hyperintense lesion on magnetic resonance imaging (MRI) after Week 8 compared to the Week 8 MRI scan.
Time Frame: Baseline up to 4 years
Population: First Enrollment Cohort ITT population. Treatment efficacy was measured for this First Enrollment Cohort. Number analyzed per timepoint are unique number of participants out of all the participants who were assessed at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage of participants
  Week 24: number analyzed (Participants) | 646
  Week 24 | 95.98 [94.20 to 97.23]
  Week 48: number analyzed (Participants) | 590
  Week 48 | 88.94 [86.30 to 91.09]
  Week 72: number analyzed (Participants) | 549
  Week 72 | 83.94 [80.92 to 86.52]
  Week 96: number analyzed (Participants) | 517
  Week 96 | 80.38 [77.14 to 83.21]
  Week 120: number analyzed (Participants) | 488
  Week 120 | 77.38 [73.99 to 80.39]
  Week 144: number analyzed (Participants) | 463
  Week 144 | 75.76 [72.28 to 78.86]
  Week 168: number analyzed (Participants) | 436
  Week 168 | 72.79 [69.18 to 76.05]
  Week 192: number analyzed (Participants) | 340
  Week 192 | 70.67 [66.97 to 74.04]

21. Primary Outcome: Percentage of Participants Without Relapse
Description: Relapse is defined as occurrence of new or worsening neurological symptoms attributable to MS, as determined using EDSS/FSS assessment.
Time Frame: Baseline up to 4 years
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage of Participants
  Week 24: number analyzed (Participants) | 661
  Week 24 | 98.52 [97.26 to 99.20]
  Week 48: number analyzed (Participants) | 649
  Week 48 | 97.91 [96.50 to 98.76]
  Week 72: number analyzed (Participants) | 631
  Week 72 | 96.25 [94.49 to 97.45]
  Week 96: number analyzed (Participants) | 610
  Week 96 | 95.32 [93.41 to 96.69]
  Week 120: number analyzed (Participants) | 593
  Week 120 | 93.90 [91.78 to 95.49]
  Week 144: number analyzed (Participants) | 570
  Week 144 | 93.09 [90.85 to 94.79]
  Week 168: number analyzed (Participants) | 554
  Week 168 | 92.43 [90.10 to 94.23]
  Week 192: number analyzed (Participants) | 439
  Week 192 | 91.56 [89.12 to 93.48]

22. Primary Outcome: Annualized Relapse Rate
Description: Relapse is defined as occurrence of new or worsening neurological symptoms attributable to MS, as determined using EDSS/FSS assessment. The adjusted annualized relapse rate is reported which is:
  Adjusted by age at disease diagnosis, Baseline EDSS, Presence of T1 Gd-enhanced lesion at screening and Presence of relapses in the last year prior to enrollment. Log-transformed exposure time is included as an offset variable.
  The report contains data up to week 192 of the treatment period of each individual participant.
Time Frame: Baseline up to 4 years
Population: First Enrollment Cohort ITT population. Treatment efficacy was measured for this First Enrollment Cohort.
Measure: Number (95% Confidence Interval); unit: events per participant per year
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
events per participant per year | 0.02 [0.015 to 0.027]

23. Primary Outcome: Sub Study: Number of Participants With IRRs Occurring During or Within 24 Hours Following the First Infusion After Randomization to the Shorter Infusion Substudy
Time Frame: Week 24 through Week 144
Population: ITT Population included all randomized participants in shorter infusion sub study.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy - Conventional Infusion | Substudy - Shorter Infusion
Number analyzed (Participants) | 373 | 372
Participants | 101 | 107

24. Secondary Outcome: Percentage of Participants Who Are Relapse Free
Description: as for outcome 21
Time Frame: Week 192
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 624
Percentage of Participants | 92.00 [89.7 to 94.0]

25. Secondary Outcome: Percentage of Participants With No Evidence of Protocol Defined Disease Activity
Description: Protocol-defined disease activity is defined as having at least one of the following: (1). protocol defined relapse (occurrence of new or worsening neurological symptoms attributable to Multiple Sclerosis [MS], as determined using EDSS/Functional Systems Score [FSS] assessment). (2). CDP, as determined using EDSS. (3). a T1 Gd-enhanced lesion after Week 8. (4). a new and/or enlarging T2 hyperintense lesion on magnetic resonance imaging (MRI) after Week 8 compared to the Week 8 MRI scan. Event-free rate
Time Frame: Weeks 96, 144, 192
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage of Participants
  Week 96: number analyzed (Participants) | 517
  Week 96 | 80.38 [77.14 to 83.21]
  Week 144: number analyzed (Participants) | 463
  Week 144 | 75.76 [72.28 to 78.86]
  Week 192: number analyzed (Participants) | 340
  Week 192 | 70.67 [66.97 to 74.04]

26. Secondary Outcome: Percentage of Participants Without Protocol-defined Event of Evidence of Progression (NEP)
Description: NEP is defined as no progression sustained for at least 24 weeks on all of the following three components (CDP; 20 percent [%] increase from baseline in timed 25 Foot Walk Test [T25FWT]; 20% increase from baseline in timed 9 hole peg test [9HPT]). CDP will be assessed using EDSS.
Time Frame: Weeks 96, 192
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage of Participants
  Week 96: number analyzed (Participants) | 511
  Week 96 | 79.60 [76.33 to 82.48]
  Week 192: number analyzed (Participants) | 325
  Week 192 | 69.16 [65.40 to 72.60]

27. Secondary Outcome: Percentage of Participants With no Evidence of Progression Sustained for At Least 24 Weeks and no Active Disease (NEPAD)
Description: NEPAD is defined as no progression on all of the three components of NEP (CDP, T25FWT, 9HPT), no new relapse and no enlarging or new T2 or T1 Gd-enhancing lesion. CDP will be assessed using EDSS. Relapse is defined as occurrence of new or worsening neurological symptoms attributable to MS, as determined using EDSS/FSS assessment.
Time Frame: Weeks 96, 192
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage of Participants
  Week 96: number analyzed (Participants) | 451
  Week 96 | 70.29 [66.65 to 73.62]
  Week 192: number analyzed (Participants) | 277
  Week 192 | 58.89 [54.96 to 62.60]

28. Secondary Outcome: Secondary: Change From Baseline in Multiple Sclerosis Functional Composite Score (MSFC) Total
Description: MSFC combines the following: Timed 25 Foot Walk Test [T25FWT] for leg function &ambulation measured in seconds (sec). The longer it takes to walk, higher the score indicating deterioration; 9 Hole Peg Test [9HPT] for arm & handf unction measured in sec. Higher score=more time taken to complete test indicating deterioration. Paced Auditory Serial Addition Test [PASAT] for cognitive function (score range: 0-60, higher score=better cognitive processing speed). MSFC composite={[Average(1/9-HPT)-Baseline Mean(1/9-HPT)/Baseline Std Dev(1/9-HPT)]+[-(Average T25FWT-Baseline Mean T25FWT)/Baseline Std-Dev T25FWT]+[(PASAT-3-BaselineMean PASAT-3)/Baseline Std Dev PASAT-3]}/ 3.0. MSFC is based on the concept that scores for these 3 dimensions are combined to create a single score to detect change over time in a group of MS patients. Higher composite score=better overall function. Lower score=worse overall function. Higher mean change in total MSFC score=functional improvement at cohort level.
Time Frame: Weeks 24, 48, 72, 96, 120, 144, 168, 192
Population: Treatment efficacy was measured for this First Enrollment Cohort ITT population. Number analyzed per timepoint are unique number of participants out of all the participants who were assessed at the specified timepoint. Different participants may have contributed data for each timepoint. As raw composite scores have been reported here, it is not possible to provide a score range for this scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
score on a scale
  Change at Week 24: number analyzed (Participants) | 595
  Change at Week 24 | 0.09 (0.67)
  Change at Week 48: number analyzed (Participants) | 601
  Change at Week 48 | 0.11 (0.54)
  Change at Week 72: number analyzed (Participants) | 588
  Change at Week 72 | 0.12 (0.45)
  Change at Week 96: number analyzed (Participants) | 566
  Change at Week 96 | 0.14 (0.53)
  Change at Week 120: number analyzed (Participants) | 511
  Change at Week 120 | 0.16 (0.61)
  Change at Week 144: number analyzed (Participants) | 513
  Change at Week 144 | 0.16 (0.48)
  Change at Week 168: number analyzed (Participants) | 498
  Change at Week 168 | 0.18 (0.56)
  Change at Week 192: number analyzed (Participants) | 492
  Change at Week 192 | 0.19 (0.72)

29. Secondary Outcome: Change From Baseline in MSFC Composite Timed 25 Foot Walk Test (T25FW) Score.
Description: The change in the mean score of T25FW is reported below. The time taken to walk 25 feet, typically measured in seconds. The longer it takes to walk, the higher score, which indicates deterioration. Lower times indicate better performance and greater mobility. Higher times indicate worse performance and greater impairment. Subsequently, the lower the mean change in the score over time, the better performance.
Time Frame: Baseline, Weeks 24, 48, 72, 96, 120, 144, 168, 192
Population: Treatment efficacy was measured for this First Enrollment Cohort ITT population. Number analyzed per timepoint are unique number of participants out of all the participants who were assessed at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
seconds
  Change at Week 24: number analyzed (Participants) | 650
  Change at Week 24 | -0.31 (6.62)
  Change at Week 48: number analyzed (Participants) | 647
  Change at Week 48 | -0.49 (6.88)
  Change at Week 72: number analyzed (Participants) | 627
  Change at Week 72 | -0.56 (6.99)
  Change at Week 96: number analyzed (Participants) | 617
  Change at Week 96 | -0.62 (6.95)
  Change at Week 120: number analyzed (Participants) | 560
  Change at Week 120 | -0.44 (7.94)
  Change at Week 144: number analyzed (Participants) | 562
  Change at Week 144 | -0.97 (6.25)
  Change at Week 168: number analyzed (Participants) | 554
  Change at Week 168 | -0.83 (6.64)
  Change at Week 192: number analyzed (Participants) | 543
  Change at Week 192 | 0.09 (9.37)

30. Secondary Outcome: Change From Baseline in MSFC Composite 9 Hole Peg Test (9HPT) Score
Description: The mean change in 9 Hole Peg Test (9HPT)-score is reported. Participants are instructed to place pegs one by one into each of nine holes arranged in a board stabilized with a plastic nonslip sheet on a solid table, and then to remove these pegs from the holes. Both the dominant and non-dominant hands are tested twice (two consecutive trials for each hand). The participants are required to complete two successful trials for each hand. The amount of time (in seconds) required to place and remove all nine pegs is recorded for each trial. The number of seconds it takes to complete the test, the higher raw scores, which indicates deterioration. The lower mean change in the score over time, the better the performance.
Time Frame: Weeks 24, 48, 72, 96, 120, 144, 168, 192
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
seconds
  Change at Week 24: number analyzed (Participants) | 650
  Change at Week 24 | -0.47 (14.44)
  Change at Week 48: number analyzed (Participants) | 648
  Change at Week 48 | -1.22 (11.54)
  Change at Week 72: number analyzed (Participants) | 628
  Change at Week 72 | -1.78 (8.09)
  Change at Week 96: number analyzed (Participants) | 618
  Change at Week 96 | -1.67 (10.91)
  Change at Week 120: number analyzed (Participants) | 551
  Change at Week 120 | -0.87 (15.21)
  Change at Week 144: number analyzed (Participants) | 560
  Change at Week 144 | -1.91 (8.70)
  Change at Week 168: number analyzed (Participants) | 555
  Change at Week 168 | -1.84 (10.68)
  Change at Week 192: number analyzed (Participants) | 544
  Change at Week 192 | -0.73 (17.55)

31. Secondary Outcome: Change From Baseline in MSFC Composite (Paced Auditory Serial Addition Test [PASAT]) Score
Description: Mean change in the Paced Auditory Serial Addition Test [PASAT] score is reported. PASAT measures cognitive function. A total of 60 single digit numbers are presented by an audiotape/CD-rom at a constant rate in every 3 seconds (PASAT-3). Participants are required to add each new number to the one immediately before it. Due to the relative complexity of this test, a practice trial with a set of 10 numbers should be performed before the original test. Participants are allowed up to 3 practice trials. Two sets of numbers (forms A & B) are developed to be used alternatively in every visit to minimize memorizing. The number of correct answers is recorded. The PASAT score ranges from 0 to 60, with higher values representing a better outcome in cognitive processing speed. Subsequently, higher values in mean changes from baseline over the study time indicate improvement in cognitive function.
Time Frame: Weeks 24, 48, 72, 96, 120, 144, 168, 192
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
score on a scale
  Change at Week 24: number analyzed (Participants) | 251
  Change at Week 24 | 4.18 (9.26)
  Change at Week 48: number analyzed (Participants) | 453
  Change at Week 48 | 5.40 (9.52)
  Change at Week 72: number analyzed (Participants) | 320
  Change at Week 72 | 6.33 (11.59)
  Change at Week 96: number analyzed (Participants) | 435
  Change at Week 96 | 7.66 (10.93)
  Change at Week 120: number analyzed (Participants) | 290
  Change at Week 120 | 7.69 (12.95)
  Change at Week 144: number analyzed (Participants) | 372
  Change at Week 144 | 8.45 (10.02)
  Change at Week 168: number analyzed (Participants) | 285
  Change at Week 168 | 8.47 (11.79)
  Change at Week 192: number analyzed (Participants) | 344
  Change at Week 192 | 9.64 (11.56)

32. Secondary Outcome: Change From Baseline in Cognitive Performance as Measured by Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) - Symbol Digits Modalities Test (SDMT)
Description: BICAMS is assessing cognitive processing speed and verbal and visual memory. SDMT assesses processing speed/working memory. The SDMT presents a series of nine symbols, each paired with a single digit in a key at the top of a standard sheet of paper. Participants are asked to voice the digit associated with each symbol as rapidly as possible for 90 sec. There is a single outcome measure - the number correct over the 90 second time span. The higher the results, the better processing speed/working memory.
Time Frame: Baseline, Weeks 48, 96, 144, 192
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: responses over 90 seconds
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 602
responses over 90 seconds
  Change at Week 48 | 2.48 (10.12)
  Change at Week 96: number analyzed (Participants) | 563
  Change at Week 96 | 1.89 (9.98)
  Change at Week 144: number analyzed (Participants) | 506
  Change at Week 144 | 3.33 (9.31)
  Change at Week 192: number analyzed (Participants) | 506
  Change at Week 192 | 4.38 (10.38)

33. Secondary Outcome: Change From Baseline in Cognitive Performance as Measured by BICAMS -California Verbal Learning Test-II (CVLT-II)
Description: BICAMS assesses cognitive processing speed and verbal and visual memory. The CLVT-II is an assessment of verbal learning and memory which measures recall and recognition scores, encoding strategies, learning rates and error types. A list learning task with 16 words from 4 semantic categories are read over a series of 5 list presentations. Recall is assessed after learning and at a 20-minute delay. The maximum possible score is 80 and a minimum is 0. A higher score indicated better recall.
Time Frame: Baseline, Weeks 48, 96, 144, 192
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 130
score on a scale
  Change at Week 48 | 2.02 (8.29)
  Change at Week 96: number analyzed (Participants) | 119
  Change at Week 96 | 2.71 (9.25)
  Change at Week 144: number analyzed (Participants) | 97
  Change at Week 144 | 3.99 (7.60)
  Change at Week 192: number analyzed (Participants) | 108
  Change at Week 192 | 4.28 (13.76)

34. Secondary Outcome: Change From Baseline in Cognitive Performance as Measured by BICAMS - Brief Visuospatial Memory Test-Revised (BVMT-R)
Description: BICAMS assesses cognitive processing speed and verbal and visual memory. BVMT-R assesses visuospatial memory. In this test, six abstract designs are presented for 10 sec. The display is removed from view and patients render the stimuli via pencil on paper manual responses. Each design receives from 0 to 2 points representing accuracy and location. There are three learning trials, and the outcome measure is the total number of points earned over the three learning trials, thus the scale range is 0-36. The higher the result, the better visual/spatial memory.
Time Frame: Baseline, Weeks 48, 96, 144, 192
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 643
points on a scale
  Baseline | 23.69 (6.44)
  Change at Week 48: number analyzed (Participants) | 587
  Change at Week 48 | -0.71 (5.31)
  Change at Week 96: number analyzed (Participants) | 566
  Change at Week 96 | 0.82 (5.68)
  Change at Week 144: number analyzed (Participants) | 489
  Change at Week 144 | 3.15 (5.37)
  Change at Week 192: number analyzed (Participants) | 489
  Change at Week 192 | 1.06 (7.09)

35. Secondary Outcome: Total Number of T1 Gd-Enhancing Lesions as Detected by Brain MRI
Description: Number of Lesions are categorized as followed: 1, 2, 3, >1, >3
Time Frame: Weeks 24, 48, 96, 144, 192
Population: ITT population
Measure: Number; unit: Number of Lesions
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Number of Lesions
  Week 24 Number of Lesions 0: number analyzed (Participants) | 667
  Week 24 Number of Lesions 0 | 659
  Week 24 Number of Lesions 1: number analyzed (Participants) | 667
  Week 24 Number of Lesions 1 | 6
  Week 24 Number of Lesions 2: number analyzed (Participants) | 667
  Week 24 Number of Lesions 2 | 2
  Week 24 Number of Lesions >1: number analyzed (Participants) | 667
  Week 24 Number of Lesions >1 | 2
  Week 48 Number of Lesions 0: number analyzed (Participants) | 657
  Week 48 Number of Lesions 0 | 650
  Week 48 Number of Lesions 1: number analyzed (Participants) | 657
  Week 48 Number of Lesions 1 | 7
  Week 96 Number of Lesions 0: number analyzed (Participants) | 657
  Week 96 Number of Lesions 0 | 629
  Week 96 Number of Lesions 1 | 1
  Week 144 Number of Lesions 0: number analyzed (Participants) | 569
  Week 144 Number of Lesions 0 | 567
  Week 144 Number of Lesions 1: number analyzed (Participants) | 569
  Week 144 Number of Lesions 1 | 1
  Week 144 Number of Lesions 3: number analyzed (Participants) | 569
  Week 144 Number of Lesions 3 | 1
  Week 144 Number of Lesions >1: number analyzed (Participants) | 569
  Week 144 Number of Lesions >1 | 1
  Week 192 Number of Lesions 0: number analyzed (Participants) | 546
  Week 192 Number of Lesions 0 | 545
  Week 192 Number of Lesions 1: number analyzed (Participants) | 546
  Week 192 Number of Lesions 1 | 1

36. Secondary Outcome: Total Number of New and/or Enlarging T2 Lesion as Detected by Brain MRI
Description: Number of Lesions are categorized as followed: 1, 2, 3, >1
Time Frame: Baseline, Weeks 24, 48, 96, 144, 192
Population: ITT Population
Measure: Number; unit: Number of Lesions
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Number of Lesions
  Week 24 Number of Lesions 0: number analyzed (Participants) | 667
  Week 24 Number of Lesions 0 | 651
  Week 24 Number of Lesions 1: number analyzed (Participants) | 667
  Week 24 Number of Lesions 1 | 13
  Week 24 Number of Lesions 2: number analyzed (Participants) | 667
  Week 24 Number of Lesions 2 | 3
  Week 24 Number of Lesions >1: number analyzed (Participants) | 667
  Week 24 Number of Lesions >1 | 3
  Week 48 Number of Lesions 0: number analyzed (Participants) | 660
  Week 48 Number of Lesions 0 | 644
  Week 48 Number of Lesions 1: number analyzed (Participants) | 660
  Week 48 Number of Lesions 1 | 11
  Week 48 Number of Lesions 2: number analyzed (Participants) | 660
  Week 48 Number of Lesions 2 | 3
  Week 48 Number of Lesions 3: number analyzed (Participants) | 660
  Week 48 Number of Lesions 3 | 2
  Week 48 Number of Lesions >1: number analyzed (Participants) | 660
  Week 48 Number of Lesions >1 | 5
  Week 96 Number of Lesions 0: number analyzed (Participants) | 633
  Week 96 Number of Lesions 0 | 624
  Week 96 Number of Lesions 1: number analyzed (Participants) | 633
  Week 96 Number of Lesions 1 | 8
  Week 96 Number of Lesions 2: number analyzed (Participants) | 633
  Week 96 Number of Lesions 2 | 1
  Week 96 Number of Lesions >1: number analyzed (Participants) | 633
  Week 96 Number of Lesions >1 | 1
  Week 144 Number of Lesions 0: number analyzed (Participants) | 572
  Week 144 Number of Lesions 0 | 564
  Week 144 Number of Lesions 1: number analyzed (Participants) | 572
  Week 144 Number of Lesions 1 | 6
  Week 144 Number of Lesions 2: number analyzed (Participants) | 572
  Week 144 Number of Lesions 2 | 1
  Week 144 Number of Lesions 3: number analyzed (Participants) | 572
  Week 144 Number of Lesions 3 | 1
  Week 144 Number of Lesions >1: number analyzed (Participants) | 572
  Week 144 Number of Lesions >1 | 2
  Week 192 Number of Lesions 0: number analyzed (Participants) | 551
  Week 192 Number of Lesions 0 | 546
  Week 192 Number of Lesions 1: number analyzed (Participants) | 551
  Week 192 Number of Lesions 1 | 4
  Week 192 Number of Lesions 2: number analyzed (Participants) | 551
  Week 192 Number of Lesions 2 | 1
  Week 192 Number of Lesions >1: number analyzed (Participants) | 551
  Week 192 Number of Lesions >1 | 1

37. Secondary Outcome: Change From Baseline in Total T1 Hypointense Lesion Volume as Detected by Brain MRI
Time Frame: Baseline, Weeks 48, 96, 144, 192
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Micro Liter
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Micro Liter
  Week 48: number analyzed (Participants) | 651
  Week 48 | -310.63 (708.07)
  Week 96: number analyzed (Participants) | 624
  Week 96 | -405.61 (755.99)
  Week 144: number analyzed (Participants) | 566
  Week 144 | -359.76 (761.84)
  Week 192: number analyzed (Participants) | 548
  Week 192 | -307.64 (797.87)

38. Secondary Outcome: Total Number of Fluid-Attenuated Inversion-Recovery (FLAIR) Lesion as Detected by Brain MRI
Description: Fluid-Attenuated Inversion-Recovery (FLAIR) Lesion as Detected by Brain MRI was measured for its volumes.
Time Frame: Baseline, Weeks 8, 24, 48, 96, 144, 192
Population: First Enrollment Cohort ITT population. Treatment efficacy was measured for this First Enrollment Cohort.
Measure: Number; unit: Number of Lesions
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Number of Lesions
  Baseline Week 8 0: number analyzed (Participants) | 639
  Baseline Week 8 0 | 633
  Baseline Week 8 1: number analyzed (Participants) | 639
  Baseline Week 8 1 | 6
  Week 24 0: number analyzed (Participants) | 641
  Week 24 0 | 635
  Week 24 1: number analyzed (Participants) | 641
  Week 24 1 | 6
  Week 48 0: number analyzed (Participants) | 637
  Week 48 0 | 631
  Week 48 1: number analyzed (Participants) | 637
  Week 48 1 | 6
  Week 96 0: number analyzed (Participants) | 618
  Week 96 0 | 611
  Week 96 1: number analyzed (Participants) | 618
  Week 96 1 | 7
  Week 144 0: number analyzed (Participants) | 555
  Week 144 0 | 550
  Week 144 1: number analyzed (Participants) | 555
  Week 144 1 | 5
  Week 192 0: number analyzed (Participants) | 535
  Week 192 0 | 530
  Week 192 1: number analyzed (Participants) | 535
  Week 192 1 | 5

39. Secondary Outcome: Change From Baseline in Brain Volume as Detected by Brain MRI
Description: Percentage change from Normalized brain volume in cm3 (cubic centimeter)values are reported
Time Frame: From Baseline to Weeks 24, 48, 96, 144, 192
Population: First Enrollment Cohort ITT population. Treatment efficacy was measured for this First Enrollment Cohort.
Measure: Mean (Standard Deviation); unit: Percentage Change in Volume (cm3)
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage Change in Volume (cm3)
  Week 24: number analyzed (Participants) | 420
  Week 24 | -0.189 (0.564)
  Week 48: number analyzed (Participants) | 404
  Week 48 | -0.479 (0.733)
  Week 96: number analyzed (Participants) | 352
  Week 96 | -0.909 (0.930)
  Week 144: number analyzed (Participants) | 301
  Week 144 | -1.283 (1.156)
  Week 192: number analyzed (Participants) | 266
  Week 192 | -1.535 (1.311)

40. Secondary Outcome: Percentage of Participants Without Treatment Discontinuation
Time Frame: Baseline up to 4 years
Population: First Enrollment Cohort ITT population. Treatment efficacy was measured for this First Enrollment Cohort.
Measure: Number (95% Confidence Interval); unit: Percentage %
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Percentage %
  Week 24: number analyzed (Participants) | 671
  Week 24 | 98.97 [97.85 to 99.51]
  Week 48: number analyzed (Participants) | 661
  Week 48 | 97.49 [96.00 to 98.45]
  Week 72: number analyzed (Participants) | 652
  Week 72 | 96.02 [94.25 to 97.25]
  Week 96: number analyzed (Participants) | 635
  Week 96 | 93.51 [91.38 to 95.13]
  Week 120: number analyzed (Participants) | 625
  Week 120 | 92.04 [89.73 to 93.84]
  Week 144: number analyzed (Participants) | 605
  Week 144 | 89.23 [86.65 to 91.34]
  Week 168: number analyzed (Participants) | 589
  Week 168 | 87.17 [84.41 to 89.47]
  Week 192: number analyzed (Participants) | 464
  Week 192 | 83.85 [80.85 to 86.42]

41. Secondary Outcome: Employment Status: Work Productivity and Activity Impairment Questionnaire (WAPI) Score
Description: WPAI scale measures impact of health problems on work productivity and regular activities: Absenteeism (Work Time Missed) measuring % of work time missed due to health issues; Presenteeism:Calculated as the percentage of impairment while working due to health problems. Overall Work Impairment:Calculated by combining absenteeism and presenteeism using the formula:Overall Work Impairment=Absenteeism+(1-Absenteeism)×Presenteeism Overall Work Impairment=Absenteeism+(1-Absenteeism)×Presenteeism This formula accounts for both the time missed and the reduced productivity while at work.
  Activity Impairment: Calculated as the percentage of impairment in regular activities outside of work. Range: Each component is scored as 0%-100%). Higher % indicate greater impairment and worse outcomes.
Time Frame: Baseline, Weeks 24, 48, 96, 120, 144, 192
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: WAPI Sub-Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
WAPI Sub-Score
  Work productivity Baseline: number analyzed (Participants) | 369
  Work productivity Baseline | 26.33 (31.84)
  Work productivity Week 24: number analyzed (Participants) | 401
  Work productivity Week 24 | 17.65 (25.04)
  Work productivity Week 48: number analyzed (Participants) | 404
  Work productivity Week 48 | 18.83 (25.92)
  Work productivity Week 96: number analyzed (Participants) | 420
  Work productivity Week 96 | 16.46 (23.10)
  Work productivity Week 144: number analyzed (Participants) | 368
  Work productivity Week 144 | 16.78 (23.85)
  Work productivity Week 192: number analyzed (Participants) | 369
  Work productivity Week 192 | 15.80 (22.25)
  Activity Impairment Baseline: number analyzed (Participants) | 640
  Activity Impairment Baseline | 23.23 (24.79)
  Activity Impairment Week 24: number analyzed (Participants) | 634
  Activity Impairment Week 24 | 18.09 (22.15)
  Presenteeism Week 48: number analyzed (Participants) | 635
  Presenteeism Week 48 | 18.85 (23.37)
  Activity Impairment Week 96: number analyzed (Participants) | 605
  Activity Impairment Week 96 | 17.79 (22.92)
  Activity Impairment Week 144: number analyzed (Participants) | 563
  Activity Impairment Week 144 | 17.80 (23.74)
  Activity Impairment Week 192: number analyzed (Participants) | 521
  Activity Impairment Week 192 | 18.18 (23.25)

42. Secondary Outcome: SymptoMScreen Composite Score
Description: The SMSS consists of 12 items which are assessed on a seven-point Likert scale that ranges from 0 (not at all affected) to 6 (total limitation) [7]. The total score ranges from 0 to 72, with higher scores indicating more severe symptom endorsement.
Time Frame: Baseline, Weeks 24, 48, 96, 144, 192
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Change in SymptoMScreen Composite Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Change in SymptoMScreen Composite Score
  Week 24: number analyzed (Participants) | 651
  Week 24 | -0.1 (0.9)
  Week 48: number analyzed (Participants) | 648
  Week 48 | -0.1 (1.0)
  Week 96: number analyzed (Participants) | 621
  Week 96 | 0.0 (1.1)
  Week 144: number analyzed (Participants) | 568
  Week 144 | 0.0 (1.1)
  Week 192: number analyzed (Participants) | 538
  Week 192 | 0.0 (1.1)

43. Secondary Outcome: Quality of Life: Multiple Sclerosis Impact Scale (MSIS)-29 Questionnaire Score
Description: The 29-item Multiple Sclerosis Impact Scale (MSIS-29) is a questionnaire to examine the impact of multiple sclerosis (MS) on physical and psychological functioning from a patient's perspective, which includes 29 items self-reported measures associated with a physical scale and 9 items with a psychological scale. MSIS-29 scales are generated by summing items and it's ranging from 29-145'. The higher total MSIS-29 scores indicate a greater degree of disability. The mean change in MSIS-29 scores from baseline is reported. The decreasing values in the mean change from baseline indicate functional improvement from patients' perspective
Time Frame: Baseline, Weeks 24, 48, 96, 144, 192
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Change in MSIS-29 Mean Score
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 678
Change in MSIS-29 Mean Score
  Week 24: number analyzed (Participants) | 656
  Week 24 | -2.43 (12.13)
  Week 48: number analyzed (Participants) | 650
  Week 48 | -2.15 (13.04)
  Week 96: number analyzed (Participants) | 627
  Week 96 | -1.26 (14.31)
  Week 144: number analyzed (Participants) | 571
  Week 144 | -0.73 (14.83)
  Week 192: number analyzed (Participants) | 543
  Week 192 | -0.63 (16.04)

44. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Baseline up to 4 years
Population: Safety and ITT populations
Measure: Number; unit: Percentage of Participants
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 1225
Percentage of Participants
  Adverse Events | 95.8
  Serious Adverse Events | 15.0

45. Secondary Outcome: Substudy: Number of Participants With IRR Overall and by Dose at Randomization
Time Frame: From Week 24 to Week 144
Population: ITT Population included all randomized participants in shorter infusion sub study. Number analyzed is the number of participants who received an infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy - Conventional Infusion | Substudy - Shorter Infusion
Number analyzed (Participants) | 373 | 372
Participants
  All Randomized Doses (Overall) | 155 | 172
  1st Randomized Dose | 101 | 107
  2nd Randomized Dose: number analyzed (Participants) | 367 | 355
  2nd Randomized Dose | 84 | 96
  3rd Randomized Dose: number analyzed (Participants) | 305 | 300
  3rd Randomized Dose | 62 | 82
  4th Randomized Dose: number analyzed (Participants) | 147 | 136
  4th Randomized Dose | 14 | 17
  5th Randomized Dose: number analyzed (Participants) | 23 | 21
  5th Randomized Dose | 1 | 3
  6th Randomized Dose: number analyzed (Participants) | 6 | 4
  6th Randomized Dose | 0 | 0

46. Secondary Outcome: Substudy: Severity of IRRs
Description: The number of participants with IRRs by most extreme intensity were reported (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 =life-threatening, grade 5 = fatal). Multiple IRRs in one participant are counted only once at the most extreme (highest) intensity observed.
Time Frame: From Week 24 to Week 144
Population: ITT Population included all randomized participants in shorter infusion sub study. Number analyzed is the number of participants with IRR.
Measure: Count of Participants; unit: Participants
Arm/Group | Substudy - Conventional Infusion | Substudy - Shorter Infusion
Number analyzed (Participants) | 373 | 372
Participants
  Grade 1 (Mild) | 88 | 92
  Grade 2 (Moderate) | 66 | 76
  Grade 3 (Severe) | 1 | 4
  Grade 4 (Life-Threatening) | 0 | 0
  Grade 5 (Fatal) | 0 | 0

47. Secondary Outcome: Substudy: Number of IRR Symptoms
Time Frame: From Week 24 to Week 144
Population: ITT Population included all randomized participants in shorter infusion sub study. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with an infusion.
Measure: Number; unit: symptoms
Arm/Group | Substudy - Conventional Infusion | Substudy - Shorter Infusion
Number analyzed (Participants) | 373 | 372
symptoms | 471 | 458

48. Secondary Outcome: Substudy: IRRs Leading to Treatment Discontinuation
Time Frame: From Week 24 to Week 144
Population: ITT Population included all randomized participants in shorter infusion sub study.
Measure: Number; unit: symptoms
Arm/Group | Substudy - Conventional Infusion | Substudy - Shorter Infusion
Number analyzed (Participants) | 373 | 372
symptoms | 0 | 0

ADVERSE EVENTS:
Time Frame: Main study: Up to 4 Years Sub-study: Week 24 to Week 144
Description: Safety population included all enrolled participants who received any dose or part of a dose of ocrelizumab. Three participants from the 'Substudy - Conventional Infusion' arm received shorter infusions of ocrelizumab. Hence, these participants are represented in the 'Substudy - Shorter Infusion' arm for safety assessment.
Groups:
- Ocrelizumab: Ocrelizumab was administered IV as two 300-mg infusions on Days 1 and 15, followed by one 600-mg infusion dose every 24 weeks (+/- 14 days) for a maximum of 8 doses throughout the 192 weeks treatment period.
Arm/Group | Ocrelizumab | Substudy - Conventional Infusion | Substudy - Shorter Infusion
All-Cause Mortality (participants affected / at risk) | 13/1225 | 2/370 | 1/375
Serious Adverse Events (participants affected / at risk) | 184/1225 | 21/370 | 19/375
Other Adverse Events (participants affected / at risk) | 1110/1225 | 251/370 | 276/375
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab (N=1225) | Substudy - Conventional Infusion (N=370) | Substudy - Shorter Infusion (N=375)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
PALPITATIONS (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CRI DU CHAT SYNDROME (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
THYROID CYST (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
VISUAL IMPAIRMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 1 (4) | 1 (1) | 0 (0)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 1 (1)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0)
BILE DUCT STONE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
IMMUNE RECONSTITUTION INFLAMMATORY SYNDROME (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 5 (5) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 23 (23) | 2 (2) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 17 (18) | 0 (0) | 2 (2)
EPIDIDYMITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
FALLOPIAN TUBE ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GENITAL HERPES (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
HEPATITIS A (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MENINGITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MENINGITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
ORCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PENILE ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
PERITONSILLAR ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 8 (8) | 0 (0) | 1 (1)
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
RENAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SUBACUTE ENDOCARDITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
TYPHOID FEVER (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 5 (5) | 0 (0) | 2 (2)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VAGINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VARICELLA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 6 (7) | 0 (0) | 1 (1)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
CAPILLARY PERMEABILITY INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1) | 1 (1) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
INTRADUCTAL PAPILLOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
INVASIVE DUCTAL BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
PAPILLARY THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DYSTONIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 9 (9) | 0 (0) | 0 (0)
NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
RADICULOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SEIZURE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ABORTION (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 1 (1) | 0 (0)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
HAEMORRHAGE IN PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
DEPRESSIVE SYMPTOM (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0)
MAJOR DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (4) | 0 (0) | 0 (0)
POST-TRAUMATIC STRESS DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
SOMATIC SYMPTOM DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 2 (3) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 1 (2) | 0 (0) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
UTERINE POLYP (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
VULVOVAGINAL PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
NASAL TURBINATE HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 4 (4) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
PHLEBITIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab (N=1225) | Substudy - Conventional Infusion (N=370) | Substudy - Shorter Infusion (N=375)
DIARRHOEA (Gastrointestinal disorders) | 91 (116) | 18 (18) | 9 (10)
NAUSEA (Gastrointestinal disorders) | 87 (109) | 8 (11) | 10 (10)
FATIGUE (General disorders) | 201 (274) | 28 (32) | 28 (29)
PYREXIA (General disorders) | 98 (139) | 7 (12) | 8 (9)
BRONCHITIS (Infections and infestations) | 62 (84) | 6 (6) | 8 (11)
COVID-19 (Infections and infestations) | 291 (344) | 14 (14) | 13 (13)
INFLUENZA (Infections and infestations) | 96 (119) | 8 (8) | 9 (9)
NASOPHARYNGITIS (Infections and infestations) | 320 (646) | 58 (81) | 50 (70)
ORAL HERPES (Infections and infestations) | 63 (142) | 5 (18) | 9 (11)
PHARYNGITIS (Infections and infestations) | 63 (81) | 8 (8) | 9 (9)
SINUSITIS (Infections and infestations) | 109 (144) | 8 (12) | 13 (14)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 196 (301) | 28 (34) | 35 (41)
URINARY TRACT INFECTION (Infections and infestations) | 184 (319) | 20 (30) | 24 (30)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 674 (1930) | 154 (297) | 172 (350)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 132 (169) | 17 (21) | 15 (20)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 115 (147) | 12 (15) | 14 (16)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 68 (76) | 11 (12) | 11 (12)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 133 (172) | 18 (24) | 14 (14)
DIZZINESS (Nervous system disorders) | 88 (102) | 12 (12) | 10 (10)
HEADACHE (Nervous system disorders) | 295 (639) | 46 (80) | 37 (50)
HYPOAESTHESIA (Nervous system disorders) | 91 (113) | 17 (20) | 11 (14)
PARAESTHESIA (Nervous system disorders) | 98 (124) | 20 (25) | 15 (17)
ANXIETY (Psychiatric disorders) | 62 (69) | 10 (11) | 8 (8)
DEPRESSION (Psychiatric disorders) | 75 (88) | 11 (13) | 11 (14)
INSOMNIA (Psychiatric disorders) | 81 (85) | 12 (12) | 9 (9)
COUGH (Respiratory, thoracic and mediastinal disorders) | 126 (160) | 13 (15) | 18 (19)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 113 (156) | 7 (7) | 9 (13)
RASH (Skin and subcutaneous tissue disorders) | 84 (109) | 9 (9) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/10/NCT03085810/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT03085810/SAP_001.pdf